CLINICAL TRIAL: NCT00267332
Title: A Randomized Double-Blinded, Placebo Controlled, Crossover Trial Examining the Effectiveness of Modafinil in Opioid Induced Sedation
Brief Title: Modafinil in Opioid Induced Sedation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: J0502
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cancer; Pain
Keywords: Sedation; Pain; modafinil; opioids
MeSH Terms: conditions — Neoplasms; Pain | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
* The primary objective of this study is to evaluate the efficacy of modafinil in the treatment of opioid induced sedation as measured by the Epworth Sleepiness Scale (ESS).
* The secondary objective is to estimate the frequency and severity of toxicity associated with Modafinil (400mg) in patients with opioid induced sedation.

DETAILED DESCRIPTION:
Sedation is a common side effect of opioid analgesics. In patients where this remains a dose limiting toxicity, stimulants (caffeine, methylphenidate, ephedrine, amphetamine) have been the primary class of agents used to counteract sedation. Modafinil is a novel stimulant that is FDA approved for the treatment of narcolepsy and has a very different side effect profile than traditional stimulants. The potential role of this agent in the treatment of opioid induced sedation remains undefined. This study, which utilizes a prospective, randomized, blinded, cross-over design, will collect daily information on sedation (Epworth Sleepiness Scale), pain, opioid consumption, and adverse effects in 90 patients suffering from opioid induced sedation within the Johns Hopkins Medical Institutions.

ELIGIBILITY:
Inclusion Criteria:

* Epworth Sleepiness Scale > 10
* Etiology of sleepiness is attributed only to opioids
* Patient must have been taking an opioid for more than 2 weeks or have been on a non-escalating dose of opioids for at least 1 week
* Patient must be able to give written informed consent
* Age >18 years

Exclusion Criteria:

* Hypersensitivity to modafinil
* Mini-Mental Status Exam (MMSE) < 25/30
* Renal impairment (calculated creatinine clearance < 40)
* Hepatic dysfunction (total bilirubin > 1.8, AST > 75IU/l, ALT > 100IU/l, prothrombin time > 40%
* Known history of cardiovascular disease (i.e., left ventricular hypertrophy, ischemic ECG changes, chest pain, arrhythmia, mitral valve prolapse, recent myocardial infarction, unstable angina, uncontrolled hypertension)
* Woman who are pregnant, breast-feeding or on hormonal contraception
* Patients taking tricyclic antidepressants, CNS stimulants, hormonal contraceptives or drugs that are inhibitors or inducers of CYP 3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Sedation
Pain

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Grossman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States